CLINICAL TRIAL: NCT00685009
Title: Women's Health Initiative Memory Study
Brief Title: The Women's Health Initiative Memory Study (The WHIMS Study)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 548; N01WH44221 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Dementia Syndromes
Keywords: Cognition; Memory; Hormone Therapy
MeSH Terms: interventions — Estrogen Replacement Therapy; Estrogens, Conjugated (USP); Estrogens; Prempro

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Women from the Women's Health Initiative study taking estrogen hormone therapy
  Interventions: Drug: Estrogen hormone therapy
- 2: Women from the WHI study taking estrogen plus progesterone hormone therapy
  Interventions: Drug: Estrogen plus progesterone hormone therapy
- 3: Women from the WHI study taking placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estrogen hormone therapy — Estrogen pill daily
  Other Names: Premarin
  Groups: 1
Drug: Estrogen plus progesterone hormone therapy — Estrogen plus progesterone hormone therapy pill (Prempro) daily
  Other Names: Prempro
  Groups: 2
Drug: Placebo — Placebo pill daily
  Groups: 3

SUMMARY:
Excessive memory decline or dementia affects an increasing number of women as they become older. The frequency of dementia doubles every 5 years beginning at age 60, making the discovery of ways to prevent or slow the disease imperative. Previous studies have indicated that changes in memory may be associated with the female hormonal decline that occurs after menopause, but more research is needed to establish the link between menopause and poorer memory function. It is believed that taking the female hormones estrogen and/or progesterone may help improve women's health by protecting against memory decline. This study will evaluate the effects of female hormone replacement therapy (HRT) on the development and progression of memory loss in older women enrolled in the Women's Health Initiative (WHI) study.

DETAILED DESCRIPTION:
Diseases of the memory, including dementia and Alzheimer's disease, are a primary health concern of the aging population. In just the last 30 years, the number of Americans diagnosed with memory diseases has doubled. The beginning signs and symptoms of Alzheimer's and dementia include mild forgetfulness, confusion, and disorientation with time and place. As the diseases advance, people often experience difficulty in carrying out normal activities, recognizing family and friends, and eventually speaking and comprehending. Early identification and treatment for dementia and Alzheimer's may help prevent and slow the progression of symptoms, but the most beneficial means of treatment is still unknown. Previous studies have suggested a link between menopause and reduced memory function in women, possibly attributed to the dramatic decline in the levels of the female hormones estrogen and progesterone. HRT in postmenopausal women may help to curb memory loss and reduce risk of developing memory-related diseases. This study will evaluate the effects of female HRT on the development and progression of memory loss in older women enrolled in the WHI study.

Participants in this study will be drawn from the WHI study and will have previously been assigned to HRT with estrogen, HRT with estrogen plus progesterone, or placebo. During this study, participants will continue to take their assigned treatments from the WHI study.

Participation will last up to 6 years. All participants will undergo baseline memory and thinking tests, including a mood assessment and tasks measuring memory and other brain functions. Study staff will conduct a telephone interview with a close family member or friend. Some participants may additionally undergo a 45-minute interview with a clinician, a blood draw, and a computerized tomography (CT) scan. All participants will repeat the baseline memory and thinking tests once annually for 6 years, and some participants will repeat the interview, blood draw, and CT scan at these annual visits as well.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Women's Health Initiative - Hormone Therapy Trial
* Aged 65 - 79 years of age at time of enrollment

Ages: 65 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will include participants from the hormone therapy trial of the WHI study.
Sampling Method: Non-Probability Sample
Enrollment: 7525 (Actual)
Dates: Start 1996-01; Primary Completion 1997-09 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
All-cause dementia | Measured annually for 6 years

SECONDARY OUTCOMES:
Mild cognitive impairment | Measured annually for 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Sally A. Shumaker, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Shumaker SA, Reboussin BA, Espeland MA, Rapp SR, McBee WL, Dailey M, Bowen D, Terrell T, Jones BN. The Women's Health Initiative Memory Study (WHIMS): a trial of the effect of estrogen therapy in preventing and slowing the progression of dementia. Control Clin Trials. 1998 Dec;19(6):604-21. doi: 10.1016/s0197-2456(98)00038-5. PMID 9875839
- [Derived] Harris WS, Tintle NL, Manson JE, Metherel AH, Robinson JG. Effects of menopausal hormone therapy on erythrocyte n-3 and n-6 PUFA concentrations in the Women's Health Initiative randomized trial. Am J Clin Nutr. 2021 Jun 1;113(6):1700-1706. doi: 10.1093/ajcn/nqaa443. PMID 33710263
- [Derived] Lo K, Liu Q, Madsen T, Rapp S, Chen JC, Neuhouser M, Shadyab A, Pal L, Lin X, Shumaker S, Manson J, Feng YQ, Liu S. Relations of magnesium intake to cognitive impairment and dementia among participants in the Women's Health Initiative Memory Study: a prospective cohort study. BMJ Open. 2019 Nov 3;9(11):e030052. doi: 10.1136/bmjopen-2019-030052. PMID 31685499
- [Derived] Haring B, Wu C, Coker LH, Seth A, Snetselaar L, Manson JE, Rossouw JE, Wassertheil-Smoller S. Hypertension, Dietary Sodium, and Cognitive Decline: Results From the Women's Health Initiative Memory Study. Am J Hypertens. 2016 Feb;29(2):202-16. doi: 10.1093/ajh/hpv081. Epub 2015 Jul 1. PMID 26137952
- [Derived] Espeland MA, Pettinger M, Falkner KL, Shumaker SA, Limacher M, Thomas F, Weaver KE, Stefanick ML, McQuellon C, Hunt JR, Johnson KC. Demographic and health factors associated with enrollment in posttrial studies: the Women's Health Initiative Hormone Therapy Trials. Clin Trials. 2013;10(3):463-72. doi: 10.1177/1740774513477931. Epub 2013 Mar 12. PMID 23480899